CLINICAL TRIAL: NCT04699708
Title: Carbon -Di-Oxide Monitoring During Neonatal STAbilization at Delivery
Brief Title: Co2 Monitoring at Preterm Delivery-Observational Study
Acronym: COSTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 291372
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Resuscitation
Keywords: Carbon dioxide monitoring; Preterm; Resuscitation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants ≤ 32 weeks: All preterm infants ≤ 32 weeks born in two study centers receiving resuscitative measures at the time of birth either in the form of face mask ventilation or intubation.
  Interventions: Device: Carbon dioxide monitoring

INTERVENTIONS:
Device: Carbon dioxide monitoring — Blinded recording of CO2 during preterm resuscitation.

SUMMARY:
CO2 data, serving as a proxy marker for tidal volume, might enable titration of tidal volume/pressure thereby providing optimal ventilation during neonatal resuscitation.

Currently there is insufficient data on Co2 levels for preterm babies requiring resuscitation. This study involves monitoring of CO2 during preterm stabilisation.

DETAILED DESCRIPTION:
Measurement of exhaled CO2 in the delivery room is feasible, but clinical benefits of during neonatal transition have not been studied. Volume ventilation in the Neonatal unit has been shown to improve outcomes such BPD or death. Despite the proven benefits of volume ventilation in the neonatal unit volume guided resuscitation at birth remains an unproven and under-studied technique.

CO2 data, serving as a proxy marker for tidal volume, might enable titration of tidal volume/pressure thereby providing optimal ventilation during neonatal resuscitation. Currently there is insufficient data on Co2 levels for preterm babies requiring resuscitation. This data would help in finding out optimal resuscitation strategies (Pressures/volume, frequency of breaths) rather than providing the same for all infants throughout the process of resuscitation and would help us in better interpretation Co2 levels in the future resuscitation.

Investigators aim to study the impact of various clinical (Gestation, Birth weight, need for intubation/bag-mask ventilation) and resuscitative factors (use of inflation pressures, ventilation pressures, frequency of breaths, face mask ventilation, intubation) on CO2 during preterm stabilisation.

ELIGIBILITY:
Inclusion Criteria:

1. All preterm infants ≤ 32 weeks born at the study centres.
2. Needing resuscitative measures at the time of birth either in the form of face mask ventilation or intubation.

Exclusion Criteria:

1. Preterm infants below the threshold of viability as determined by the study team.
2. Major congenital or chromosomal abnormality (including congenital heart disease, Diaphragmatic hernia, congenital pulmonary airway malformations).
3. Severe oligohydramnios (Amniotic fluid index <5 or deep vertical pool≤2).

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm infants ≤ 32 weeks born in two study centers receiving resuscitative measures at the time of birth either in the form of face mask ventilation or intubation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Factors influencing carbon dioxide levels during preterm resuscitation | 1 year
  To study the impact/correlation of various clinical factors (Gestation, Birth weight, need for intubation/bag-mask ventilation, surfactant administration, delayed cord clamping) and resuscitative factors (use of inflation pressures, ventilation pressures, frequency of breaths, face mask ventilation, intubation) on carbon dioxide measurements using MASIMO NOMOLINE capnography during preterm stabilisation.

SECONDARY OUTCOMES:
Correlation of Co2 with other parameters | 1 year
  Correlation between oxygen saturation, CO2 and pulse rate.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - James Cook University Hospital, Middlesbrough, Stockton ON TEES
  - Imran Ahmed, Sunderland

IPD SHARING:
Plan to Share IPD: Undecided